CLINICAL TRIAL: NCT05189457
Title: A Phase IIA Study of Sequential ("First Strike, Second Strike") Therapies, Modeled on Evolutionary Dynamics of Anthropocene Extinctions, for High Risk Metastatic Castration Sensitive Prostate Cancer
Brief Title: First Strike, Second Strike Therapies for High Risk Metastatic Castration Sensitive Prostate Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: BeiGene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-21139
Record Dates: First submitted 2021-12-29; First posted 2022-01-12 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: Prostate Cancer; Stage IV Prostate Cancer
Keywords: Prostate; Metastatic prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Gonadotropin-Releasing Hormone; Leuprolide; Triptorelin Pamoate; relugolix; acetyl-2-naphthylalanyl-3-chlorophenylalanyl-1-oxohexadecyl-seryl-4-aminophenylalanyl(hydroorotyl)-4-aminophenylalanyl(carbamoyl)-leucyl-ILys-prolyl-alaninamide; abiraterone; enzalutamide; Docetaxel; tislelizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- First Strike then Second Strike (Experimental): The first part of the study treatment or "first strike" involves 12-18 weeks of combined therapy with LHRH analog and one of the new hormonal agents (NHAs). Participants will complete the "first strike" at week 13 if their PSA has reduced >90%; otherwise they will complete a total of 18 weeks of therapy. The second part of the treatment or "second strike" involves 4 cycles docetaxel and LHRH analog. The "second strike" will start immediately after the "first strike". MRI guided prostate biopsy will be performed after "second strike". For patients with positive prostate biopsy or detectable PSA, the "second strike" will be consolidated with 4-6 additional cycles of docetaxel plus 6 doses of tislelizumab at 200 mg, given IV once every 3 weeks. For patients with undetectable PSA at year 3 from study enrollment, LHRH analog can be discontinued.
  Interventions: Drug: Luteinizing Hormone Releasing Hormone; Drug: New Hormonal Agent; Drug: Docetaxel; Drug: Tislelizumab

INTERVENTIONS:
Drug: Luteinizing Hormone Releasing Hormone — During the first strike, LHRH will be administered for 12 to 18 weeks. During the second strike, participants will receive 4 cycles of LHRH
  Other Names: Leuprolide; Triptorelin; Goserslin; Relugolix; Degarelix
Drug: New Hormonal Agent — During the first strike, if Abiraterone is chosen 1000mg of Abiraterone will be taken orally. If Enzalutamide is used, 160 mg will be taken orally every 24 hours.
  Other Names: Abiraterone; Enzalutamide
Drug: Docetaxel — During the second strike, participants will receive 4 cycles of Docetaxel at 75mg/m2 given intravenously at day 1 of ever 21 days. For participants with positive prostate biopsy or detectable PSA, the "second strike" will receive 2 additional cycles of docetaxel.
Drug: Tislelizumab — During the second strike, participants will receive 6 doses of Tislelizumab at 200 mg, given intravenously once every 3 weeks.
  Other Names: BGB-A317

SUMMARY:
The goal of this clinical research is to find if sequential therapy with combined androgen deprivation or hormonal therapy with luteinizing hormone release hormone (LHRH) analog plus a new hormonal agent (abiraterone, enzalutamide, or apalutamide) followed by chemohormonal therapy with docetaxel and LHRH analog would improve the outcome of high risk metastatic/stage IV prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy proven prostate cancer and the diagnosis can be established through either prostate biopsy or biopsy of a metastatic lesion. High risk mCSPC is defined as having 2 of the 3 risk factors: a Gleason score of 8 or more, at least 3 bone metastases, and the presence of measurable visceral metastasis.
* ECOG performance status of 0-1
* No androgen deprivation therapy (ADT) with LHRH analogue monotherapy for more than 12 weeks after the diagnosis of metastatic prostate cancer. Prior ADT in the non-metastatic setting is allowed if it was given > 2 years prior to the diagnosis of metastatic prostate cancer and a reduction of PSA is documented after initiating ADT in the metastatic setting.
* Agreeable to prostate biopsy after completing "second strike".
* Adequate organ function with absolute neutrophil count > 1000/l, Hb > 10 g/dl, Platelet > 100,000/l, Creatinine and liver enzymes within 1.5 folds of upper limits of normal
* No uncontrolled arrhythmia; participants with h/o myocardial infarction or history of congestive heart failure, need to have estimated left ventricle ejection fraction above 40% either on echocardiogram or MUGA scan within 6 months of study enrollment.
* All men who are sexually active with a female partner of childbearing potential treated or enrolled on this protocol must agree to use highly effective barrier contraception prior to the study, for the duration of study participation, and for 7 months after last dose of tislelizumab administration.
* Ability to understand and the willingness to sign a written informed consent document or have a legally authorized representative sign on the participants behalf. Stated willingness to comply with all study procedures and availability for the duration of the study
* - Inclusion of minorities: Men of all races and ethnic groups who met the above inclusion criteria are eligible for this trial.

Exclusion Criteria:

* Prior treatments with TAK-700/Orteronel, abiraterone, darolutamide, apalutamide or enzalutamide for more than eight weeks.
* Any previous treatment with a PD-1 or PD-L1 inhibitor
* Documented brain metastases
* Prior prostatectomy
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to docetaxel (including any drugs formulated with polysorbate 80), or LHRH analogue (e.g., leuprolide, triptorelin, goserelin acetate, degarelix)
* Treatment with any investigational compound within 30 days prior to the first dose of study drugs
* Diagnosis or treatment for another systemic malignancy within 2 years before the first dose of study drugs, or previously diagnosed with another malignancy & have any evidence of residual disease. Participants with non-melanoma skin cancer or carcinoma in situ of any type are not excluded if they have undergone complete resection.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Participants with delayed healing of wounds, ulcers, and/or bone fractures
* Known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome. HIV-positive participants on combination antiretroviral therapy are ineligible because of the potential for tislelizumab to be less clinically active in this population.
* Active or prior documented autoimmune or inflammatory disorders, including inflammatory bowel disease (e.g., Crohn's disease), systemic lupus erythematosus, Sarcoidosis syndrome, Grave's disease, rheumatoid arthritis, hypophysitis, uveitis, with the following exceptions: • Vitiligo or alopecia • Hypothyroidism stable on hormone replacement • Chronic skin condition that does not require systemic therapy • Celiac disease controlled by diet alone • Participants with inactive disease in the last 5 years may be included.
* Active infection including tuberculosis, hepatitis B (known positive HBV surface antigen [HBsAg]), or hepatitis C (HCV). Participants with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HBsAg) are eligible. Participants with positive HCV antibody are eligible if polymerase chain reaction is negative for HCV RNA.
* Concurrent or prior use of immunosuppressive medication within 14 days before the first dose of study chemoimmunotherapy, with the following exceptions: premedication for docetaxel with 8 mg oral dexamethasone approximately 12 hr, 8 hr and 1 hr prior to each docetaxel administration; intranasal, inhaled, topical steroids, or local steroid injections (e.g., intraarticular injection); systemic corticosteroids at physiologic doses not exceeding 10mg/day of prednisone or its equivalent; steroids as premedication for hypersensitivity reactions (e.g., premedication for iodinated contrast allergy before CT scan)
* History of severe hypersensitivity reactions to chimeric or humanized antibodies or fusion proteins
* History of interstitial lung disease, non-infectious pneumonitis or uncontrolled diseases including pulmonary fibrosis, acute lung diseases, etc.
* Was administered a live vaccine ≤ 4 weeks before first dose of tislelizumab NOTE:Seasonal vaccines for influenza and COVID-19 vaccines are generally inactivated vaccines and are allowed. Intranasal vaccines are live vaccines and are not allowed.
* Inability to comply with protocol requirements
* Inclusion of minorities: Men of all races and ethnic groups who met the above exclusion criteria are eligible for this trial.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2022-01-25 (Actual); Primary Completion 2027-07-15 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | Up to 36 months
  Overall survival will be from initiation of first strike until failure or death from any cause.

SECONDARY OUTCOMES:
PSA <0.2 nanogram per milliliter (ng/ml) rate at 6 months | At 6 months
  Investigators will measure the PSA <0.2 nanogram per milliliter (ng/ml) at 6 months from the initiation of the first strike
PSA <0.2 nanogram per milliliter (ng/ml) rate at 12 months | At 12 months
  Investigators will measure the PSA <0.2 nanogram per milliliter (ng/ml) at 12 months from the initiation of the first strike
PSA <0.2 nanogram per milliliter (ng/ml) rate at 36 months | At 36 months
  Investigators will measure the PSA <0.2 nanogram per milliliter (ng/ml) at 36 months from the initiation of the first strike
PSA Progression | Up to 36 months
  Time to PSA progression from the initiation of "first strike"
Radiographic Progression | At 36 months
  Investigators will measure the radiographic progression free survival rate at 36 months from the initiation of "first strike"

OTHER OUTCOMES:
Comparison of Standard Uptake Values (SUV) | Up to 9 months
  Investigators will track the changes on F18 (Posluma or Pylarify) PSMA PET scan after first and second strikes compared to baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Jingsong Zhang, MD, PhD, Principal Investigator — Moffitt Cancer Center
Locations (1):
- Moffitt Cancer Center, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Moffitt Cancer Center Clinical Trial Web Search — https://moffitt.org/clinical-trials-research/clinical-trials/